CLINICAL TRIAL: NCT06453291
Title: Innovative Approaches in Managing Chronic Low Back Pain: A Comparative Assessment of Clinical Techniques
Brief Title: Assessment of Different Clinical Techniques to Treat Patients With Chronic Low Back Pain
Acronym: CLBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iffat Anwar Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAMC002
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: CLBP; Neuromodulation; PRP
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen; Diagnosis-Related Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy Group (Experimental): * Intervention: Participants will receive standard treatment for CLBP, including NSAIDs and physical therapy.
  * Frequency: Daily NSAID use as prescribed, physical therapy sessions twice a week
  Interventions: Drug: NSAIDs (Nonsteroidal Anti-Inflammatory Drugs):; Procedure: Standard Physical Therapy
- Neuromodulation + PRP Therapy Group (Experimental): * Intervention: Participants will undergo neuromodulation via the DRG and receive PRP injections.
  * Frequency: Neuromodulation sessions once a week for the first month, followed by monthly maintenance sessions if needed. PRP injections will be administered once a week for the first three weeks.
  Interventions: Procedure: Neuromodulation via Dorsal Root Ganglion (DRG):; Procedure: Platelet-Rich-Plasma Therapy

INTERVENTIONS:
Drug: NSAIDs (Nonsteroidal Anti-Inflammatory Drugs): — Objective: To reduce pain and inflammation associated with chronic low back pain.
  Medications: Ibuprofen, Naproxen, or Diclofenac.
  Dosage:
  Ibuprofen: 400-600 mg every 6-8 hours as needed. Naproxen: 250-500 mg twice daily as needed. Diclofenac: 50 mg three times daily as needed. Administration: Oral tablets. Duration: Daily use as prescribed, for the duration of the study. Monitoring: Regular follow-up visits to monitor pain levels, side effects, and adherence.
  Other Names: Ibuprofen; Naproxin
  Arms: Conventional Therapy Group
Procedure: Standard Physical Therapy — Objective: To improve mobility, strength, and reduce pain.
  Techniques:
  Stretching exercises. Strengthening exercises for core and back muscles. Manual therapy techniques. Postural training. Frequency: Twice a week sessions. Duration: 45-60 minutes per session. Monitoring: Progress will be assessed during each session and adjusted as necessary
  Other Names: Muscle strengthening
  Arms: Conventional Therapy Group
Procedure: Neuromodulation via Dorsal Root Ganglion (DRG): — Objective: To modulate excitatory pathways and reduce pain through targeted stimulation.
  Procedure:
  Placement of electrodes near the DRG. Application of pulsed radiofrequency (RF) at 42°C for 3-20 minutes.
  Frequency:
  Initial treatment: Once a week for the first month. Maintenance: Monthly sessions if needed. Duration: Each session lasts approximately 30-45 minutes. Monitoring: Pain levels and functional improvement will be assessed before and after each session.
  Other Names: Pulsed RF
  Arms: Neuromodulation + PRP Therapy Group
Procedure: Platelet-Rich-Plasma Therapy — Objective: To promote healing and reduce inflammation through the application of concentrated platelets.
  Procedure:
  Blood draw from the patient. Centrifugation to separate platelets. Injection of PRP into the affected area of the lower back.
  Frequency:
  Initial treatment: Once a week for the first three weeks. Follow-up: Additional injections may be given based on patient response and clinical judgment.
  Duration: Each session lasts approximately 30-45 minutes. Monitoring: Pain levels, inflammation markers, and functional improvement will be assessed before and after each injection.
  Other Names: platelet concentrates
  Arms: Neuromodulation + PRP Therapy Group

SUMMARY:
This clinical trial aims to assess the effectiveness of different clinical techniques in treating patients with chronic low back pain (CLBP). Two test groups will be included: one receiving conventional therapy (NSAIDs and other physical therapy techniques) and the other receiving a combination of neuromodulation and platelet-rich plasma (PRP) therapy. Chronic pain, persisting for more than three months, inhibits natural pathways like GABA and promotes excitatory pathways, leading to increased inflammation. The study hypothesizes that neuromodulation via the dorsal root ganglion (DRG) and PRP therapy will provide superior pain relief and functional improvement compared to conventional therapy.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) affects millions of individuals worldwide, significantly impacting quality of life and productivity. Traditional treatments often involve NSAIDs and physical therapy, but these methods sometimes fail to provide adequate relief. Chronic pain is characterized by prolonged activation of the central and peripheral nervous systems, resulting in sensitization and increased pain perception.

The current study will evaluate two treatment modalities:

1. Conventional Therapy: This includes the use of nonsteroidal anti-inflammatory drugs (NSAIDs) and other standard physical therapy techniques.
2. Neuromodulation + PRP Therapy: Neuromodulation is performed via the DRG to modulate excitatory pathways, with medial sensory nerves being desensitized at 42°C for 3-20 minutes. PRP therapy involves the injection of concentrated platelets to promote healing and reduce inflammation.

The study will provide valuable insights into the comparative effectiveness of these treatments, potentially guiding future therapeutic strategies for CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-60 years.
* Diagnosed with chronic low back pain persisting for more than three months.
* Willingness to participate and comply with study procedures.
* Ability to provide informed consent.

Exclusion Criteria:

* Comorbidities.
* Contagious and Non-Contagious Infections
* Known hypersensitivity to study interventions.
* Presence of severe psychiatric disorders.
* Pregnancy or breastfeeding.
* Participation in another clinical trial within the last 30 days.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 0 Weeks
  Improvement in the Visual Analog Scale (VAS)
Visual Analog Scale (VAS) | 2 Weeks
  Improvement in the Visual Analog Scale (VAS)
Visual Analog Scale (VAS) | 3 Months
  Improvement in the Visual Analog Scale (VAS)
Visual Analog Scale (VAS) | 6 Months
  Improvement in the Visual Analog Scale (VAS)
Visual Analog Scale (VAS) | 12 Months
  Improvement in the Visual Analog Scale (VAS)
Oswestry Disability Index (ODI) | 0 weeks
  Improvement in the Oswestry Disability Index (ODI)
Oswestry Disability Index (ODI) | 2 weeks
  Improvement in the Oswestry Disability Index (ODI)
Oswestry Disability Index (ODI) | 3 Months
  Improvement in the Oswestry Disability Index (ODI)
Oswestry Disability Index (ODI) | 6 Months
  Improvement in the Oswestry Disability Index (ODI)
Oswestry Disability Index (ODI) | 12 Months
  Improvement in the Oswestry Disability Index (ODI)
Hospital Anxiety Depression (HAD) | 0 Weeks
  Improvement in the Hospital Anxiety Depression (HAD)
Hospital Anxiety Depression (HAD) | 2 Weeks
  Improvement in the Hospital Anxiety Depression (HAD)
Hospital Anxiety Depression (HAD) | 3 Months
  Improvement in the Hospital Anxiety Depression (HAD)
Hospital Anxiety Depression (HAD) | 6 Months
  Improvement in the Hospital Anxiety Depression (HAD)
Hospital Anxiety Depression (HAD) | 12 Months
  Improvement in the Hospital Anxiety Depression (HAD)

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad Anwar, MBBS, DOM, Principal Investigator — Iffat Anwar Medical Complex, Lahore
Locations (1):
- Iffat Anwar Medical Complex, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Ho KY, Gwee KA, Cheng YK, Yoon KH, Hee HT, Omar AR. Nonsteroidal anti-inflammatory drugs in chronic pain: implications of new data for clinical practice. J Pain Res. 2018 Sep 20;11:1937-1948. doi: 10.2147/JPR.S168188. eCollection 2018. PMID 30288088
- [Background] Deer T, Pope J, Hayek S, Narouze S, Patil P, Foreman R, Sharan A, Levy R. Neurostimulation for the treatment of axial back pain: a review of mechanisms, techniques, outcomes, and future advances. Neuromodulation. 2014 Oct;17 Suppl 2:52-68. doi: 10.1111/j.1525-1403.2012.00530.x. PMID 25395117
- [Background] Sundman EA, Cole BJ, Karas V, Della Valle C, Tetreault MW, Mohammed HO, Fortier LA. The anti-inflammatory and matrix restorative mechanisms of platelet-rich plasma in osteoarthritis. Am J Sports Med. 2014 Jan;42(1):35-41. doi: 10.1177/0363546513507766. Epub 2013 Nov 5. PMID 24192391